CLINICAL TRIAL: NCT01076894
Title: Analgesia and Pulmonary Function After Thoracic Surgery: is an Intercostal Nerve Block Plus Intravenous Morphine as Effective as Epidural Anesthesia? A Prospective Randomized Clinical Study.
Brief Title: Thoracotomy: Intercostal Nerve Block Versus Epidural Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Department of Anesthesiology, University Clinic Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDA-ICB 198/06
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Thoracotomy
Keywords: pain; thoracotomy; pulmonary function; epidural anesthesia; intercostal nerve block
MeSH Terms: conditions — Pain | interventions — Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- epidural anesthesia (Active Comparator)
  Interventions: Procedure: epidural anesthesia
- intercostal anesthesia (Active Comparator)
  Interventions: Procedure: intercostal anesthesia

INTERVENTIONS:
Procedure: epidural anesthesia — In the epidural group prior to the induction of general anesthesia, a thoracic epidural catheter will be was placed at the level of the TH6-TH8. 8 ml ropivacaine 1% were administered through the epidural catheter. EDA is aimed at a sensory block level from TH2 to TH10.
  Arms: epidural anesthesia
Procedure: intercostal anesthesia — In the intercostal group, before chest closure, each 4 ml ropivacaine 0.75 % will be injected by the surgeon under direct vision into the proximal intercostal space at the level of the thoracotomy and two spaces above and below as well as 5 ml ropivacaine 0,75 % at the thoracic drainage tube exits
  Arms: intercostal anesthesia

SUMMARY:
Postoperative pain and consecutive reduction of pulmonary function after thoracic surgery still is a major clinical problem and challenge in anesthesia. Thoracic epidural anesthesia is commonly considered to be the "gold standard" for postoperative pain control and restoration of pulmonary function after thoracic surgery.

Thus, the aim of the present study is to investigate whether an intercostal nerve block with ropivacaine plus intravenous PCA with morphine is as effective as thoracic epidural anesthesia with respect to postoperative pain control and pulmonary

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective pulmonary surgery, including pneumonectomy, bilobectomy, lobectomy, typical and atypical segmentectomy, via a lateral or posterolateral thoracotomy without chest-wall resection

Exclusion Criteria:

* age<18 yr
* any contraindication to epidural anaesthesia, intercostal nerve block or the use of ropivacaine, morphine, metamizol or diclofenac
* lack of patient's cooperation
* any type of chronic painful condition or current opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Pain at rest and on coughing after thoracic surgery | Pain during the first four postoperative days

SECONDARY OUTCOMES:
pulmonary function (peak expiratory flow rate) after thoracic surgery | first four postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Georgieff, Prof., Study Chair — Department for Anesthesiology University Clinic Ulm
Locations (1):
- Universtity Clinic Ulm, Ulm, Germany